CLINICAL TRIAL: NCT06845462
Title: Application of Artificial Intelligence Algorithm Based on CT Imaging for Muscle Parameter Measurement in the Diagnosis of Sarcopenia
Brief Title: Application of Artificial Intelligence Algorithm Based on CT Imaging for Muscle Parameter Measurement
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Yaomin Hu, Administrative Director of Geriatrics Department, RenJi Hospital
Other Study IDs: LY2023-150-A
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Deep Learning; Sarcopenia; Computed Tomography; Body Composition
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To establish an artificial intelligence model for automated diagnosis of sarcopenia based on CT imaging

DETAILED DESCRIPTION:
With the accelerating aging process, the early identification and diagnosis of sarcopenia, along with the effective prevention of its adverse outcomes, have become a focal point in medical research. However, current methods for assessing and diagnosing sarcopenia still face significant limitations, making the development of more efficient and accurate techniques for muscle mass evaluation an urgent clinical need. Although CT is considered as the most promising method for assessing muscle mass, its practical application is hindered by factors such as reliance on physician expertise and time-consuming procedures, limiting its widespread clinical adoption. In light of these challenges, this study aims to develop an artificial intelligence model for fully automated muscle mass measurement based on abdominal CT imaging and to validate its application value in assisting the diagnosis of sarcopenia.

ELIGIBILITY:
Inclusion criteria：

1. The population undergoing BIA and abdominal CT examinations;
2. Can cooperate to complete human body composition analysis, grip strength measurement, 6m walking time measurement, and questionnaire survey.

Exclusion criteria：

1. Age<18 years old;
2. Existence of abdominal wall edema;
3. History of spinal surgery or vertebral fractures, or vertebral tumor lesions;
4. History of neuromuscular disorders.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 960 inpatients in the geriatric department of Renji Hospital, 20 patients from Ruijin Hospital affiliated to Shanghai Jiaotong University School of Medicine, 20 patients from The First Affiliated Hospital of Zhejiang Medical University, 50 patients from The First Affiliated Hospital of Wenzhou Medical University, and 30 patients from Huangshan People's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1080 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
To automatedly and precisely quantify three-dimensional muscle volume and fat volume. | 2020-2023
  To achieve an automated and precise quantification of three-dimensional muscle volume and fat volume at the L3 vertebral region by deep learning.
To establish an artificial intelligence model for diagnosis of sarcopenia. | 2020-2023
  The validation of artificial intelligence models can assist in the diagnosis of sarcopenia.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiaotong University School of Medicine, Renji Hospital Ethics Committee, Shanghai, Shanghai Municipality, China